CLINICAL TRIAL: NCT02196493
Title: An Open Label Trial of Azithromycin in Chronic Productive Cough
Acronym: AZCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13031; 2013-002938-20 (EudraCT Number)
Record Dates: First submitted 2014-07-10; First posted 2014-07-22 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Cough
Keywords: Productive; Cough; Bronchitis; Azithromycin
MeSH Terms: conditions — Chronic Cough; Cough; Bronchitis | interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Azithromycin (Experimental): 250mg azithromycin three times weekly for 12 weeks
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — 250mg azithromycin three times per week for 12 weeks
  Other Names: Zithromax

SUMMARY:
We have noticed a group of patients presenting with a longstanding wet cough which has often been treated as asthma. The cough is productive of sputum which frequently contains bacteria, but does not resolve with standard antibiotic treatment.

A very similar cough is seen in subjects who smoke, have exposure to airbourne dusts or chemicals or have a condition known as bronchiectasis, but these problems have already been excluded.

We have found that prolonged treatment with an antibiotic called azithromycin is very effective but using azithromycin in this way is not licensed and there is currently no trial evidence to support its use.

This research will evaluate the clinical benefit of low dose azithromycin to determine if this is an effective and safe treatment for these patients. It will also involve a detailed investigation of these patients to determine whether they have enough in common to believe we are describing a new condition.

DETAILED DESCRIPTION:
We and others have observed a cohort of patients, mainly referred with either poorly controlled asthma despite high dose treatment or suspected bronchiectasis, who give a history of chronic (often 3 months or more) productive cough which improves with antibiotic treatment but quickly relapses. Most deny wheeze and on examination there are often transmitted sounds from mucus in the large airways but no expiratory wheeze typical of asthma. Investigations including spirometry, bronchial challenges, chest X-ray, screen for immunodeficiency and high resolution CT (HRCT) scan exclude recognised causes of productive cough but sputum culture is often positive for Haemophilus influenzae although sometimes demonstrates normal respiratory flora despite being markedly purulent.

Due to their efficacy in cystic fibrosis and bronchiectasis we have empirically tried treatment with low dose macrolide antibiotics over 3-6 months often with dramatic benefit. This is however an unproven and unlicensed indication which needs to be more thoroughly evaluated.

The key objective of the study is to determine if 12 weeks treatment of patients with chronic productive cough with low dose azithromycin is both effective and safe.

The secondary objectives of the study are to describe the clinical and pathological features of a cohort of patients who present with chronic productive cough (with no evidence of bronchiectasis, smoking-related chronic bronchitis or immunodeficiency) to determine if these are sufficiently similar to justify a new diagnostic label.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Male or female
* Non-smokers for 10 years and <20 pack year equivalents in total
* Persistent productive cough for > 3 months in duration
* Use of effective contraception Acceptable contraceptive methods include: established use of oral, injected or implanted hormonal methods; placement of an intrauterine device (IUD) or intrauterine system (IUS); condom or occlusive cap (diaphragm or cervical/vault caps) with spermicide; true abstinence (when this is in line with the preferred and usual lifestyle of the participant); or vasectomised partner.

Exclusion Criteria:

* History of obvious inhaled irritant exposure
* Evidence of primary or secondary immunodeficiency.
* Clinically important bronchiectasis on HRCT scan
* Prolonged QT interval on ECG or significant cardiac pathology prior to commencing azithromycin
* Abnormal LFT's (greater than 2x upper limit of normal)
* Hypersensitivity to azithromycin or any macrolide/ketolide antibiotic
* Pregnancy or intent to become pregnant during course of study
* Contra-indication to bronchoscopy (as per British Thoracic Society Guidelines)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in cough on the Leicester Cough Questionnaire (LCQ) score at week 12 | 12 weeks after treatment started

SECONDARY OUTCOMES:
Change from baseline in sputum colour (as per previously validated commercially available graded sputum colour chart) at week 12 | 12 weeks after treatment started
Change from baseline in exhaled nitric oxide level (ppm) at week 24 | 12 weeks after treatment started
Change from baseline in FEV1 (ml) at week 24 | 12 weeks after treatment started
Change from baseline in sputum volume (ml) at week 12 | 12 weeks after treatment started

CONTACTS AND LOCATIONS:
Overall Officials: Tim Harrison, MD, FRCP, Principal Investigator — University of Nottingham
Locations (1):
- Respiratory Research Unit, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martin MJ, Lee H, Clayton C, Pointon K, Soomro I, Shaw DE, Harrison TW. Idiopathic chronic productive cough and response to open-label macrolide therapy: An observational study. Respirology. 2019 Jun;24(6):558-565. doi: 10.1111/resp.13483. Epub 2019 Feb 5. PMID 30722097